CLINICAL TRIAL: NCT00822237
Title: Safety, Tolerability, and Immunogenicity of VARIVAX (2007 Commercial VZV Bulk Process) Administered Concomitantly With M-M-R II in Healthy Children 12-to-23 Months of Age
Brief Title: Study to Test the Safety and Immunogenicity of VARIVAX (2007 Process) (Study V210-057) (Completed)
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: V210-057; 2009_510
Record Dates: First submitted 2009-01-09; First posted 2009-01-14 (Estimated); Results first posted 2011-04-21 (Estimated); Last update posted 2017-04-12 (Actual); Status verified 2017-03

CONDITIONS: Varicella
MeSH Terms: conditions — Chickenpox | interventions — Herpes Zoster Vaccine; Measles-Mumps-Rubella Vaccine

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- VARIVAX 2007 process + M-M-R II (Experimental)
  Interventions: Biological: Varicella Virus Vaccine Live (2007 Process) (Oka/Merck); Biological: Measles, Mumps, and Rubella Virus Vaccine Live (MMR)
- VARIVAX 1999 process + M-M-R II (Active Comparator)
  Interventions: Biological: Comparator: Varicella Virus Vaccine Live (1999 Process) (Oka/Merck); Biological: Measles, Mumps, and Rubella Virus Vaccine Live (MMR)

INTERVENTIONS:
Biological: Varicella Virus Vaccine Live (2007 Process) (Oka/Merck) — VARIVAX (2007 process) in two 0.5 mL doses by injection ~6 weeks apart
  Arms: VARIVAX 2007 process + M-M-R II
Biological: Comparator: Varicella Virus Vaccine Live (1999 Process) (Oka/Merck) — VARIVAX (1999 process) in two 0.5 mL doses by injection ~6 weeks apart
  Arms: VARIVAX 1999 process + M-M-R II
Biological: Measles, Mumps, and Rubella Virus Vaccine Live (MMR) — M-M-R II in two 0.5 mL doses by injection ~6 weeks apart

SUMMARY:
This study will test the safety, tolerability, and immunogenicity of VARIVAX manufactured with the 2007 commercial Varicella-Zoster Virus (VZV) bulk process when concomitantly administered with M-M-R II in healthy children.

DETAILED DESCRIPTION:
This treatment has been approved for sale to the public.

ELIGIBILITY:
Inclusion Criteria:

* Subject is in good health based on medical history
* Subject has no history of measles, mumps, rubella, chickenpox, or shingles

Exclusion Criteria:

* Subject has previously received measles, mumps, rubella, and/or varicella vaccine either alone or in combination
* Subject has history of immune disorders
* Subject has been exposed to chickenpox/shingles, measles, mumps, rubella or varicella within 4 weeks of study start
* Subject has received an inactivated vaccine within 14 days of first dose of study vaccine
* Subject has received a live vaccine within 30 days of first dose of study vaccine
* Subject has received a blood transfusion or blood-derived products within 3 months of receiving study vaccine
* Subject has had a fever within 72 hours of study start

Ages: 12 Months to 23 Months | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 598 (Actual)
Dates: Start 2009-01; Primary Completion 2009-10 (Actual); Study Completion 2009-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Monitor, Study Director — Merck Sharp & Dohme LLC

IPD SHARING:
Plan to Share IPD: Yes
http://www.merck.com/clinical-trials/pdf/Merck%20Procedure%20on%20Clinical%20Trial%20Data%20Access%20Final_Updated%20July_9_2014.pdf
  http://engagezone.msd.com/ds_documentation.php

RESULTS

PARTICIPANT FLOW:
Groups:
- VARIVAX 2007 Process + M-M-R II: VARIVAX (2007 process) in two 0.5 mL doses by injection ~6 weeks apart
  M-M-R II (Measles, Mumps, and Rubella Virus Vaccine Live) in two 0.5 mL doses by injection ~6 weeks apart
- VARIVAX 1999 Process + M-M-R II: VARIVAX (1999 process) in two 0.5 mL doses by injection ~6 weeks apart
  M-M-R II (Measles, Mumps, and Rubella Virus Vaccine Live) in two 0.5 mL doses by injection ~6 weeks apart
Period: Dose 1 Vaccination
Arm/Group | VARIVAX 2007 Process + M-M-R II | VARIVAX 1999 Process + M-M-R II
Started | 299 (Number randomized) | 299 (Number randomized)
Completed | 274 | 273
Not Completed | 25 | 26
Not completed — Not vaccinated | 3 | 0
Not completed — Withdrawal by Subject | 13 | 14
Not completed — Lost to Follow-up | 9 | 12
Period: Dose 2 Vaccination
Arm/Group | VARIVAX 2007 Process + M-M-R II | VARIVAX 1999 Process + M-M-R II
Started | 274 (Number who received second dose) | 273 (Number who received second dose)
Completed | 270 | 262
Not Completed | 4 | 11
Not completed — Withdrawal by Subject | 2 | 2
Not completed — Lost to Follow-up | 2 | 9

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | VARIVAX 2007 Process + M-M-R II | VARIVAX 1999 Process + M-M-R II | Total
Number analyzed (Participants) | 299 | 299 | 598
Age, Continuous [Mean (Standard Deviation); unit: months] | 13.0 (1.83) | 13.0 (1.83) | 13.0 (1.83)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 158 | 138 | 296
  Male | 141 | 161 | 302

OUTCOME MEASURES:

1. Primary Outcome: Percent of Participants Who Achieved Varicella Immunogenicity After a Single Dose of VARIVAX (2007 Process).
Description: Percent of participants with varicella antibody titer ≥ 5 Glycoprotein Enzyme-Linked Immunosorbent Assay (gpELISA) units/mL in participants with baseline varicella antibody titer < 1.25 gpELISA units/mL.
  Results for the VARIVAX (1999 Process) arm are not included in this table because the primary outcome measure is for the VARIVAX (2007 Process) arm only.
Time Frame: 6 weeks following first vaccination
Population: Per protocol population
Measure: Number; unit: Percent of participants
Arm/Group | VARIVAX 2007 Process + M-M-R II
Number analyzed (Participants) | 246
Percent of participants | 96.3

ADVERSE EVENTS:
Description: Number of participants at risk for the 2007 process is the number who received the first dose.
Arm/Group | VARIVAX 2007 Process + M-M-R II | VARIVAX 1999 Process + M-M-R II
Serious Adverse Events (participants affected / at risk) | 1/296 | 1/299
Other Adverse Events (participants affected / at risk) | 189/296 | 156/299
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | VARIVAX 2007 Process + M-M-R II (N=296) | VARIVAX 1999 Process + M-M-R II (N=299)
Croup infectious (Infections and infestations) | 1 (1) | 0 (0)
Bronchial hyperreactivity (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | VARIVAX 2007 Process + M-M-R II (N=296) | VARIVAX 1999 Process + M-M-R II (N=299)
Diarrhoea (Gastrointestinal disorders) | 24 (27) | 17 (24)
Vomiting (Gastrointestinal disorders) | 20 (23) | 13 (15)
Injection site erythema (General disorders) | 67 (134) | 64 (137)
Injection site pain (General disorders) | 84 (205) | 70 (167)
Injection site swelling (General disorders) | 32 (69) | 35 (63)
Irritability (General disorders) | 27 (34) | 15 (21)
Pyrexia (General disorders) | 74 (110) | 65 (92)
Otitis media (Infections and infestations) | 31 (33) | 22 (25)
Upper respiratory tract infection (Infections and infestations) | 20 (24) | 20 (22)
Cough (Respiratory, thoracic and mediastinal disorders) | 12 (17) | 16 (18)
Dermatitis diaper (Skin and subcutaneous tissue disorders) | 21 (24) | 15 (16)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The SPONSOR must have the opportunity to review all proposed abstracts, manuscripts, or presentations regarding this study 60 days prior to submission for publication/presentation. Any information identified by the SPONSOR as confidential must be deleted prior to submission. SPONSOR review can be expedited to meet publication guidelines.